CLINICAL TRIAL: NCT05759884
Title: Efficacy Analysis of Anti-vascular Endothelial Growth Factor (VEGF) Drugs Combined With Micropulse Laser in the Treatment of Diabetic Macular Edema
Brief Title: Efficacy Analysis of Anti-VEGF Drugs Combined With Micropulse Laser in the Treatment of Diabetic Macular Edema
Acronym: VEGF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0022
Record Dates: First submitted 2023-02-08; First posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-02

CONDITIONS: Macular Edema Due to Type 2 Diabetes Mellitus
Keywords: Macular Edema
MeSH Terms: conditions — Macular Edema

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anti-VEGF combined SML therapy group (Experimental): The patients were treated with intravitreal injection of anti-VEGF drugs and SML therapy.
  Interventions: Drug: Anti-VEGF; Radiation: subthreshold micropulse laser
- anti-VEGF single therapy group (Active Comparator): Only intravitreal injection of anti-VEGF drugs was given to patients.
  Interventions: Drug: Anti-VEGF

INTERVENTIONS:
Drug: Anti-VEGF — Intravitreous injection of anti-VEGF drugs
Radiation: subthreshold micropulse laser — 577nm micropulse laser photocoagulation therapy
  Arms: anti-VEGF combined SML therapy group

SUMMARY:
The goal of this clinical trial is to clarify the efficacy of anti-vascular endothelial growth factor (anti-VEGF) drugs combined with subthreshold micropulse laser (SML) therapy on retinal function and anatomical recovery in patients with diabetic macular edema (DME). The main questions it aims to answer are:

* To clarify the efficacy of anti-VEGF drugs combined with SML therapy on retinal function and anatomical recovery in DME patients.
* To explore the changes in visual acuity and optical coherence tomography angiography (OCTA) parameters before and after the treatment of DME with anti-VEGF drugs combined with SML, and further explore the changes in morphological characteristics of retinal microvessels and the potential treatment mechanism.

Participants will randomly be given Intravitreous injection of anti-VEGF drugs or anti-VEGF drugs combined with SML therapy. All participants will be followed up for 6 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-proliferative diabetic retinopathy (NPDR) meeting diagnostic criteria: the diagnosis can be made by fundus examination, fluorescein fundus angiography (FFA) and optical coherence tomography (OCT), which meet the clinical significant macular edema (CSME) definition criteria, i.e. hard exudation within 500μm of macular fovea with adjacent retinal thickening or edema within 500μm of macular fovea. Or the thickened area of the retina was > 1 disc diameter (D) and within 1 day of the fovea of the macula.
* OCT examination showed a thickened CMT (≥200μm) without hyperplasia or scar
* Standard logarithmic visual acuity charts measure the BCVA (LogMAR) range from 0.01 to 1.0
* Control of glycosylated hemoglobin (HbA1c) ≤10% during follow-up
* Patients voluntarily participate and sign informed consent

Exclusion Criteria:

* Patients with severe corneal opacity, cataract and vitreous hemorrhage were found to be affected by OCTA examination by ophthalmic examination.
* Patients with other eye diseases or other complications during follow-up, such as glaucoma (IOP>21mmHg), high myopia (≥-6.0D), and other fundus lesions, such as retinal detachment, vitreous macular traction, preretinal membrane, ischemic macular disease, optic neuritis and other diseases involving the retina and optic nerve.
* Patients who have previously received intraocular surgery, vitreous macular traction syndrome, proliferative diabetic retinopathy (PDR) resulting in vitreous hemorrhage or local retinal detachment requiring surgical treatment, and patients with a history of eye trauma.
* History of panretinal photocoagulation within 6 months prior to treatment or local/grille photocoagulation within 3 months prior to treatment.
* History of intravitreal injection of any steroid within 6 months prior to treatment.
* Patients with serious systemic diseases, such as cardiovascular and cerebrovascular diseases or hematopoietic system, patients who have undergone intracranial surgery or intracranial space-occupying lesions, and patients with mental disorders.
* Can not cooperate with the ophthalmic examination or other reasons can not obtain the ideal OCTA image.
* Pregnant, pregnant or lactating women and patients allergic to drugs.
* Suspected or confirmed history of alcohol and drug abuse.
* Patients who are participating in clinical trials of other drugs. If one of the above meets and can be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
central macular thickness (CMT) | up to 6 months
  CMT

SECONDARY OUTCOMES:
best-corrected visual acuity (BCVA) | up to 6 months
  BCVA
superficial capillary vessel density (SVD) | up to 6 months
  The vessel density of the superficial capillary plexus level will be analyzed in the 3×3 mm OCTA scanning mode.
deep capillary vessel density (DVD) | up to 6 months
  The vessel density of the deep capillary plexus level will be analyzed in the 3×3 mm OCTA scanning mode.
foveal avascular zone (FAZ) | up to 6 months
  The area of FAZ will be evaluated on 3×3 mm OCTA image.
nonperfusion (NP) | up to 6 months
  The NP regions in the superficial and deep capillary plexuswere will be evaluated on the 3×3 mm OCTA Image by Image J software. The scores were as follows: 1 for 0~3 NP regions, 2 for 4~6 NP regions, and 3 for more than 6 NP regions.

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No